CLINICAL TRIAL: NCT01992978
Title: The Influence of Radiofrequency-assisted Hepatectomy on the Perioperative Outcomes and the Long-term Prognosis of HCC With Cirrhosis：A Prospective Randomized Controlled Trial
Brief Title: Radiofrequency-assisted Hepatectomy on the Outcomes of HCC Patients With Cirrhosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Southwest Hospital, China (Other)
Responsible Party: Principal Investigator, Li Xiaowu,MD, Dr.Xiaowu Li, Southwest Hospital, China
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SWHB2013-005
Record Dates: First submitted 2013-11-11; First posted 2013-11-25 (Estimated); Last update posted 2015-11-24 (Estimated); Status verified 2015-11

CONDITIONS: Hepatocellular Carcinoma; Cirrhosis
Keywords: radiofrequency-assisted（RF）; hepatectomy; postoperative liver injury
MeSH Terms: conditions — Carcinoma, Hepatocellular; Fibrosis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- radiofrequency-assisted resection group（RF-R) (Experimental): Radiofrequency-assisted resection: separating the tumor from liver by using the probe of radiofrequency to block the arterial and vessels before parenchymal transection.
  Interventions: Procedure: Radiofrequency-assisted Hepatectomy
- conventional liver resection group（CLR-R） (Active Comparator): Conventional liver resection group: hepatectomy only without RF assisted during parenchymal transection.Separating and dissecting the tumor with the routine clamp-crushing technical.
  Interventions: Procedure: Conventional Hepatectomy

INTERVENTIONS:
Procedure: Radiofrequency-assisted Hepatectomy — Radiofrequency-assisted resection: separating the tumor from liver by using the probe of radiofrequency to block the arterial and vessels before parenchymal transection.
  Arms: radiofrequency-assisted resection group（RF-R)
Procedure: Conventional Hepatectomy — Hepatectomy was conducted without RF assisted during parenchymal transection. Separating and dissecting the tumor with the routine clamp-crushing technical.
  Arms: conventional liver resection group（CLR-R）

SUMMARY:
Surgical resection is the most effective treatment of primary and secondary liver tumors. Technical innovations have mainly focused on minimizing bleeding during transection of the hepatic parenchyma because excessive hemorrhage and the need for blood transfusion are associated with increased postoperative morbidity and mortality. Recently,radiofrequency-assisted（RFA）hepatectomy has developed rapidly and gained widespread acceptance for the treatment of hepatocellular carcinomas（HCC），but its influence on the prognosis of HCC patients，especially for those with cirrhosis，is still controversial. Therefore, we design this prospective clinical trial to explore the effect of RFA hepatectomy versus the conventional hepatectomy on the outcomes of perioperative period and prognosis of HCC patients with cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

* Aged from 18 to 65 years , no gender restriction.
* Clinical diagnosis of resectable HCC.
* Preoperative liver function test showed Child-Pugh Class A or B.
* Indocyanine green retention at 15 minutes (ICG-15) of <30%.
* Acceptable clotting profile :platelet count > 50 x 109/L and a prolonged prothrombin time of < 5 seconds.
* Enough relative residual liver volume (%RLV) ≥ 40%.
* No tumor invasion in primary branch of portal vein, hepatic vein, or inferior vena cava.
* No other anti-tumor therapy received before the treatment.
* No metastasis in lymphnode or other organs.
* Written consent inform assigned.

Exclusion Criteria:

* Pregnancy.
* Intraoperative findings of tumor rupture，extrahepatic tumor or lymphnode metastasis.
* Tumor invasion in primary branch of portal vein, hepatic vein, or inferior vena cava.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2013-11; Primary Completion 2017-11 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Postoperative liver injury | postoperative 90 days
  The degree of postoperative hepatic injury is assessed by daily measurements of postoperative aminotransferase (AST) and alanine aminotransferase (ALT) levels, serum bilirubin levels, and prothrombin times. Each patient is followed up within postoperative 90 days.

SECONDARY OUTCOMES:
Number of Participants with Adverse Events | postoperative 90 days
  It is evaluated according to the the Clavien-Dindo Classification of surgical complications. Postoperative mortality and morbidity are measured.
Overall survival | 1,3,5-year overall survival

OTHER OUTCOMES:
Blood parameter change after operation | discharge from hospital (2 weeks)
  Blood parameter change after operation is measured by postoperative blood routine test till the hospitalization. The estimated average postoperative hospitalization ranges from 10 ot 15 days (generally 2 weeks). If the incidence of postoperative hepatic insufficiency occurred beyond hospitalization,blood routine test is also necessarily counted in.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaowu Li, MD-Ph D, Study Director — Institute of hepatobiliry surgery,Southwest hospital
Locations (1):
- Institute of Hepatobiliry surgery,Southwest Hospital, Chongqing, Chongqing Municipality, China